CLINICAL TRIAL: NCT04099979
Title: A Non-Interventional Pilot Study to Explore the Role of Gut Flora in Psoriasis
Brief Title: A Pilot Study to Explore the Role of Gut Flora in Psoriasis
Status: Withdrawn | Type: Observational
Why Stopped: Company focus shifted
Sponsor: ProgenaBiome (Other)
Responsible Party: Sponsor
Other Study IDs: PRG-011
Record Dates: First submitted 2019-09-20; First posted 2019-09-23 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Psoriasis; Psoriasis Vulgaris; Psoriasis Universalis; Psoriasis Face; Psoriasis Nail; Psoriatic Plaque; Psoriasis Diffusa; Psoriasis Punctata; Psoriasis Palmaris; Psoriasis Circinata; Psoriasis Annularis; Psoriasis Genital; Psoriasis of Scalp; Psoriasis Geographica
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool Samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Psoriasis patients: Patients who have been diagnosed with Psoriasis
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — There is no intervention for this study

SUMMARY:
This study seeks to correlate microbiome sequencing data with information provided by patients and their medical records regarding Psoriasis.

DETAILED DESCRIPTION:
The goal of this Research Study is to better understand how the genetic information in subject's microbiome correlates to the information provided in surveys and in medical records regarding Psoriasis

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent by patient
2. Male or female patients age 18 and older.
3. Diagnosis of Psoriasis based on PSAI of greater than or equal to 12 at screening

Exclusion Criteria:

1. Refusal by patient to sign informed consent form
2. Treatment with antibiotics within 2 weeks prior to screening
3. Treatment with probiotics within 6 weeks prior to screening
4. History of bariatric surgery, total colectomy with ileorectal anastomosis or proctocolectomy.
5. Postoperative stoma, ostomy, or ileoanal pouch
6. Participation in any experimental drug protocol within the past 12 weeks
7. Treatment with total parenteral nutrition
8. Any clinically significant evidence of disease that could interfere with the subject's ability to enter the trial
9. Inability of patient to adequately communicate with the investigator or their respective designee and/or comply with the requirements of the entire study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients 18 years of age or older who have been diagnoed with Psoriasis
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-03-02 (Estimated); Primary Completion 2030-03 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
Correlation of Microbiome to Psoriasis via Relative Abundance Found in Microbiome Sequencing | 1 year
  Relative abundance of bacterial classes within taxonomic phyla and, more broadly, within their domain will be analyzed by sequencing the gut microbiome. These data will then be correlated with specific Psoriasis types

SECONDARY OUTCOMES:
Validation of Sequencing Methods | 1 year
  To validate the methods used to sequence samples

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Hazan, MD, Principal Investigator — ProgenaBiome
Locations (1):
- ProgenaBiome, Ventura, California, United States

IPD SHARING:
Plan to Share IPD: Undecided
Only aggregated and deidentified data will be shared with other researchers.